CLINICAL TRIAL: NCT01202058
Title: An Observational Safety Evaluation of Patients Treated With the NEVO™ Sirolimus-eluting Coronary Stent.
Brief Title: An Observational Safety Evaluation of Patients Treated With the NEVO™ Sirolimus-eluting Coronary Stent. (NEVO II)
Acronym: NEVO II
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The NEVO™ stent will not be commercialized. Cordis decided to close the study after 1 years. This decision took the absence of safety signals into account.
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC09-01
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Atherosclerotic Coronary Artery Disease
Keywords: Coronary artery disease; Drug-eluting stents; Reservoir technology
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEVO™ SES (Experimental): Design Protocol Am3.0 - safety follow-up:
  The study population consists of 103 subjects with atherosclerotic coronary artery disease treated with the NEVO™ SES. Candidates for the initial NEVO II Study must have met ALL inclusion criteria and NO exclusion criteria.
  Design Original Protocol
  Subjects randomized to treatment with the NEVO™ Sirolimus-eluting Coronary Stent System.
  Interventions: Device: NEVO™ Sirolimus-eluting Coronary Stent System
- XIENCE V®/XIENCE PRIME™/PROMUS® (Active Comparator): Subjects randomized to treatment with the XIENCE V®/XIENCE PRIME™/PROMUS® Everolimus-eluting Coronary Stent System
  Interventions: Device: XIENCE V®/XIENCE PRIME™/PROMUS® Everolimus-eluting Coronary Stent System)

INTERVENTIONS:
Device: NEVO™ Sirolimus-eluting Coronary Stent System — Design Original Protocol
  Intervention will consist of percutaneous coronary intervention for treatment of a single or multiple coronary lesion(s) using standard coronary intervention techniques. Intervention in this arm will include treatment with the NEVO™ Sirolimus-eluting Coronary Stent System. Subjects assigned to the IVUS sub-study population will undergo intravascular ultrasound evaluation immediately post-stenting.
  Arms: NEVO™ SES
Device: XIENCE V®/XIENCE PRIME™/PROMUS® Everolimus-eluting Coronary Stent System) — Intervention will consist of percutaneous coronary intervention for treatment of a single or multiple coronary lesion(s) using standard coronary intervention techniques. Intervention in this arm will include treatment with the XIENCE V®/XIENCE PRIME™/PROMUS® Everolimus-eluting Coronary Stent System. Subjects assigned to the IVUS sub-study population will undergo intravascular ultrasound evaluation immediately post-stenting.
  Arms: XIENCE V®/XIENCE PRIME™/PROMUS®

SUMMARY:
As a result of the implementation of Protocol Am3.0, the design and objective of the NEVO II trial were changed to focus on the safety follow-up of the 103 NEVO™ subjects. Although this trial started interventional, the remainder of the study will be observational.

The objective of this prospective, observational study is to ensure the safety and the wellbeing of subjects treated with the NEVO™ SES.

DETAILED DESCRIPTION:
Restenosis remains a frequent cause of late failure after initially successful coronary angioplasty occurring in as many as 20-40% of procedures performed. Loss of luminal diameter as a result of restenosis has been attributed to three physiologic mechanisms: passive elastic recoil of the vessel, geometric vessel remodeling and neointimal hyperplasia. Coronary stents provide mechanical scaffolding that reduces restenosis by limiting the extent of elastic recoil and late vascular remodeling. Despite these improvements, the incidence of restenosis following coronary stent implantation occurs in 20-40% of cases. Restenosis following stenting is primarily a result of neointimal hyperplasia.

The methodology in interventional cardiology has historically evolved from diagnostic coronary angiography to balloon angioplasty, the use of bare metal stents, their refinement to drug-eluting stents with a durable polymer, and is now on the verge to drug-eluting stents with further developed drug delivery approaches such as the reservoir technology and the use of bioresorbable polymers. While the reservoir approach may make drug delivery more controllable, the reduction of polymer exposure to the vessel wall was designed to improve vascular healing and reduce the occurrence of undesirable side effects such as stent thrombosis especially on the long-term once the drug is completely eluted.

While to date, these are concepts validated preferably in pre-clinical studies, and only limited clinical data are available to suggest efficacy and safety of the NEVO™ SES, this study seeks to assess its clinical value in a large and unselected cohort of subjects representing real-world contemporary treatment patterns through a non-inferiority comparison with the most widely used DES today, the XIENCE V® / XIENCE PRIME™ / PROMUS® stent.

Between August and October 2010, 156 subjects were enrolled in the trial. Of the 156 subjects, 103 were treated with the NEVO™ Sirolimus-eluting Stent and 53 with the comparator. Based on a small number of acute performance observations, Cordis voluntary suspended enrollment to optimize the balloon catheter.

As a result of evolving market dynamics, and product portfolio decisions, Cordis decided in June 2011 to no longer pursue the development of NEVO™ Sirolimus-eluting coronary stents. As a result of this decision, the design and objective of the NEVO II trial were changed to allow only follow-up of the 103 NEVO™ subjects.

Since the NEVO™ SES is an investigational device; the NEVO™ subjects are being followed-up to safeguard their safety and wellbeing. The 53 subjects from the comparator arm do not need further follow-up due to the fact that they have been treated with a commercially available stent.

ELIGIBILITY:
Inclusion Criteria:

* Subject has atherosclerotic coronary artery disease with an indication for stent implantation;
* Target lesion(s) with a diameter stenosis of minimally 50% (visual estimate) OR a functional study documenting the hemodynamic relevance of the target lesion(s);
* All target lesion(s) require treatment with stents having diameters from 2.5mm to 3.5mm (visual estimate);
* Subject is ≥18 years of age;
* Subject must sign Ethics Committee approved informed consent prior to undergoing any study specific procedure;
* Subject must be willing and able to comply with specified follow-up schedule.

Exclusion Criteria:

* Planned medical procedures or concomitant disease requiring modification of DAPT regimen within 6 months of enrollment into this study;
* Women of childbearing potential without negative pregnancy test within 7 days before enrollment OR women who do not agree to remain on birth control until angiographic follow-up at 13 months if applicable OR lactating women. For women of childbearing potential, requiring an acute, non-elective procedure, a verbal confirmation of non-pregnancy and birth control is sufficient;
* Currently participating in an investigational study that has not completed the primary endpoint or that clinically interferes with the study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Twelve month composite clinical endpoint of all death, all MI and all revascularizations. | 12 months

SECONDARY OUTCOMES:
Stent thrombosis defined as definite, probable, possible and composite of definite and probable at early, late and very late time points (using ARC definition) | 60 months
Bleeding complication | 60 months
Stroke | 60 months
Device, Procedural and Lesion Success | Procedural
Composite endpoint of all death, all MI and all revascularization and its individual components | 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W. Serruys, MD, PhD, Principal Investigator — Erasmus MC - Thoraxcenter, Rotterdam, The Netherlands; Stephan Windecker, MD, PhD, Principal Investigator — Inselspital, Bern, Switzerland; Manel Sabate, MD, Principal Investigator — Hospital Universitari Clinic de Barcelona, Barcelona, Spain
Locations (3):
- Erasmus MC - Thoraxcenter, Rotterdam, Netherlands
- Hospital Universitari Clinic de Barcelona, Barcelona, Spain
- Inselspital, Bern, Switzerland